CLINICAL TRIAL: NCT03457168
Title: A Prospective, Randomized, Open-label Clinical Trial on the Effects of Intensive Versus Conventional Control of Ambulatory-determined Asleep Systolic Blood Pressure Mean on Cardiovascular, Metabolic, and Renal Disease Risks
Brief Title: Treatment of Hypertension During Sleep
Acronym: THADEUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Ramon C. Hermida, Professor and Director, Bioengineering & Chronobiology Labs., University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: THADEUS; 2017-001410-28 (EudraCT Number); 2017/470 (Registry Identifier: State Committee of Ethics in Investigation of Galicia)
Record Dates: First submitted 2018-02-21; First posted 2018-03-07 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hypertension; Hypertension, Systolic
Keywords: Sleep-time hypertension; Ambulatory blood pressure monitoring; Hypertension chronotherapy; Asleep blood pressure; Cardiovascular risk; Type 2 diabetes; Chronic kidney disease
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label (for medication treatment), two-arms, blinded-endpoint clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants unaware of their assigned randomized group. Outcomes evaluated by an independent Events Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive asleep SBP control (Active Comparator): To reduce the asleep SBP mean up to a target <110 mmHg. Treatment of elevated asleep SBP mean
  Interventions: Procedure: Treatment of elevated asleep SBP mean
- Conventional asleep SBP control (Active Comparator): To reduce the asleep SBP mean up to a target <120 mmHg. Treatment of elevated asleep SBP mean
  Interventions: Procedure: Treatment of elevated asleep SBP mean

INTERVENTIONS:
Procedure: Treatment of elevated asleep SBP mean — To reduce asleep SBP mean determined by 48h ambulatory blood pressure monitoring up to the randomly assigned target by hypertension treatment intensification when required

SUMMARY:
On the basis of new evidence on the relationship between achieved office blood pressure (BP) measurements (OBPM) and the risk of cardiovascular disease (CVD) morbidity and mortality documented in the SPRINT trial, the recent 2017 guidelines of the American College of Cardiology (ACC) and the American Heart Association (AHA) have established lower values of 130/80 mmHg for clinic systolic BP (SBP)/diastolic BP (DBP) as new diagnostic thresholds for hypertension and therapeutic targets for treatment of all individuals aged ≥18 years regardless of age, sex, or concomitant complications including presence of diabetes, chronic kidney disease (CKD), or history of past CVD event. According to these guidelines, the new proposed ambulatory BP measurment (ABPM) thresholds for diagnosis of hypertension in adults are 130/80 and 110/65 mmHg for the awake and asleep SBP/DBP means, respectively. However, the ACC/AHA guidelines do not provide any scientific evidence documenting neither the equivalence between these ABPM thresholds and the 130/80 mmHg cut-off values for OBPM nor the potential improved CVD event-free survival time of the proposed more intensive control of ambulatory BP.

Results derived from observational prospective studies consistently document that therapeutic BP targets in hypertensive individuals, i.e., persons at increased CVD risk, should be established in terms of proper control of asleep BP. To date, no prospective randomized study has ever before evaluated which should be the adequate therapeutic ABPM target for most effective reduction of CVD risk. Accordingly, the Tratamiento de Hipertensión Arterial Durante el Sueño study (THADEUS, i.e., Treatment of Hypertension During Sleep) has been designed to prospectively evaluate if "intensive control" of asleep SBP mean proposed by the new ACC/AHA guidelines (<110 mmHg) in more effective than the so far its "conventional control" (<120 mmHg) to reduce CVD morbidity and mortality in hypertensive individuals.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE OF THE STUDY.

1.1. Clinic and ambulatory blood pressure for the diagnosis of hypertension.

The diagnosis of hypertension and all clinical decisions regarding its treatment today are still mainly based only on a limited number of daytime office blood pressure (BP) measurements (OBPM) obtained in the clinic, occasionally supplemented by wake-time self-assessments at home and work. Those casual time-unspecified OBPM disregard the mostly predictable circadian variation in BP. Various circadian rhythms may also significantly affect the pharmacokinetics and pharmacodynamics, both beneficial and adverse effects, of hypertension medications, as extensively documented. Most important, numerous outcome trials and published meta-analyses substantiate the correlation between BP level and risk of target organ injury damage and cardiovascular disease (CVD) events is much stronger for parameters derived from around-the-clock ambulatory BP monitoring (ABPM) than it is for values derived from traditional daytime OBPM. ABPM is a diagnostic tool with the added advantage that allows thorough description and quantification of all aspects of the 24h BP variation.

On the basis of this substantial and indisputable evidence, several international guidelines now propose ambulatory measurements as a requirement to confirm the office diagnosis of hypertension in adults. On the contrary, other guidelines, despite recognizing greater prognostic value of ABPM than OBPM, still recommended the use of the later for diagnosis of hypertension for "historical reasons" unjustified on the light of current available scientific evidence.

1.2. Asleep BP mean as an independent prognostic marker of CVD risk.

Specific features of the ABPM-determined 24h BP pattern have been explored as biomarkers or mediators of target tissue injury and triggers of and risk factors for CVD events -- angina pectoris, myocardial infarction, cardiac arrest, sudden cardiac death, pulmonary embolism -- and cerebrovascular events -- ischemic and hemorrhagic stroke. Numerous studies consistently substantiate a strong association between the abnormal physiologic feature of blunted sleep-time relative BP decline (non-dipper/riser BP pattern) and increased incidence of fatal and non-fatal CVD events, not only in hypertensive persons, but also in normotensive individuals.27 Furthermore, various independent prospective studies demonstrate CVD events are better predicted by the asleep than awake or 24h BP means.

Overall, such prospective ABPM studies demonstrate elevated sleep-time BP constitutes a significant CVD risk factor, independent of the daytime OBPM or ambulatory awake and 24h BP means. Nonetheless, all previous investigations addressing the merit of ABPM for predicting CVD risk, except the Monitorización Ambulatoria para Predicción de Eventos Cardiovasculares study (MAPEC, i.e., Ambulatory Blood Pressure Monitoring for Prediction of Cardiovascular Events) discussed below relied upon only a single, low-reproducible study-inclusion baseline 24h ABPM assessment per participant. Lack of systematic and multiple ABPM evaluations of participants over time in all previously reported long-term follow-up studies, except MAPEC, precluded the opportunity to explore the potential reduction in CVD risk associated with modification of prognostic parameters by hypertension therapy and/or lifestyle changes, i.e., either increase of sleep-time relative BP decline towards the more normal dipper pattern or, more specifically, reduction of asleep BP mean. Incorporation of periodic (at least annual) ABPM studies of participants during follow-up, as in the MAPEC study, clearly establishes that: (i) features of the 24h BP pattern change over time; and (ii) therapeutic reduction of the asleep BP mean and increase of the sleep-time relative BP decline towards normal dipping lessen not only CVD risk but also progression towards new-onset type 2 diabetes and chronic kidney disease (CKD).

Potential reduction in CVD risk through modification of prognostic ABPM parameters by a time-specified hypertension-treatment strategy has so far been investigated only in the MAPEC study. Cox regression survival analysis of each potential prognostic BP parameter analyzed individually indicates the hazard ratio (HR) of total CVD events is greater with progressively higher sleep-time SBP mean and lower sleep-time relative SBP decline, i.e., more non-dipper/riser BP patterning. Moreover, joint analysis of the multiple BP parameters potentially capable of contributing to CVD risk finds OBPM does not independently predict CVD morbidity and mortality when the outcomes model is adjusted by the asleep BP mean (HR=1.44, 95%CI [1.30-1.60], P<0.001, per SD elevation in asleep SBP mean; HR=1.09 [0.97-1.23], P=0.123, per SD elevation in clinic SBP). The best Cox regression fully adjusted model includes only the asleep SBP mean (HR=1.43, 95%CI [1.29-1.58], P<0.001) and sleep-time relative SBP decline (HR=0.88 [0.78-0.98], P=0.023).

1.3. Asleep BP mean as a therapeutic target for CVD risk reduction.

Data from the MAPEC study, in which participants were repeatedly assessed by periodic 48h ABPM, also permitted prospective evaluation of the impact of changes in OBPM and ABPM during follow-up on CVD risk. Progressive treatment-induced lowering of the awake, asleep, and 48h BP means, but not daytime OBPM, when each variable is analyzed individually, reveals association with significant CVD risk reduction. Most importantly, Cox survival analysis with joint inclusion of asleep and awake BP means as potential predictors indicates progressive attenuation of asleep SBP mean is significantly associated with diminished CVD risk (adjusted HR=0.67 [0.55-0.81], P<0.001, per SD decrease in asleep SBP mean), while progressive lowering of awake SBP mean is not (adjusted HR=1.00 [0.86-1.18], P=0.958, per SD decrease in awake SBP mean during follow-up). Overall, the best fully adjusted time-dependent Cox regression model includes only the progressive attenuation of the asleep SBP mean (HR=0.76, 95%CI [0.68-0.85], P<0.001, per SD decrease in asleep SBP mean) and increase in the sleep-time relative SBP decline (HR=1.19 [1.01-1.39], P=0.038, per SD decrease in sleep-time relative SBP decline during follow-up). Thus, a diminished asleep, but not awake, BP mean is a highly significant independent prognostic marker of reduced CVD morbidity and mortality risk and, therefore, constitutes a novel therapeutic target for increased event-free survival.

Thus far, apart from MAPEC, the only prospective study in which participants are evaluated periodically by ABPM is the Hygia Project, a research network primarily designed to extend the use of ABPM in primary care as a requirement for the diagnosis of hypertension, evaluation of response to treatment, and individualized assessment of CVD and other risks. Presently, the Hygia Project is composed of 40 clinical sites (primary care centers) involving 292 investigators properly trained to ABPM and all study procedures. The study was designed to evaluate in the routine primary care clinical setting, among other objectives, the prognostic value of multiple ABPM-derived parameters (mainly asleep BP mean and sleep-time relative BP decline) with OBPM for the prediction of CVD morbidity and mortality, new-onset diabetes, and new-onset CKD. The investigators so far prospectively evaluated 18,078 individuals (9,769 men/8,309 women; 59.1±14.3 [mean±SD] years of age) with baseline ambulatory BP ranging from normotension to hypertension. At inclusion and at scheduled visits (mainly annually) during follow-up, ambulatory BP was evaluated for 48 consecutive hours. During the current 5.1-year median patient follow-up, 2,311 individuals had CVD events, including 1,209 experiencing the primary outcome (composite of CVD death, myocardial infarction, coronary revascularization, heart failure, and stroke). The asleep SBP mean was the most significant prognostic marker of the primary outcome (HR=1.29 [95%CI 1.22-1.35] per SD elevation, P<0.001), independent of clinic (1.03 [0.97-1.09], P=0.315) and awake SBP (1.02 [0.94-1.10], P=0.682). Most important, the progressive treatment-induced attenuation of asleep SBP was the most significant prognostic marker of event-free survival (0.75 [95%CI 0.69-0.82] per SD decrease, P<0.001), independent of changes in office (1.07 [0.97-1.17], P=0.176) or awake SBP mean (0.96 [0.85-1.08], P=0.473) during follow-up. Only the decrease in asleep SBP mean and increase in sleep-time relative SBP decline towards the more normal dipper BP pattern remained jointly and significantly associated with reduced CVD risk. There was a highly significant decrease in risk of CVD outcome with progressively lower achieved asleep SBP mean; in particular, CVD event-rate was significantly lower in participants with achieved asleep SBP mean <105 mmHg at their final evaluation than those with achieves asleep SBP mean between 105 and 120 mmHg (3.35 vs. 7.27 events per 1,000 patients/year, respectively, P<0.001; 54% CVD risk reduction in the lower achieved asleep SBP mean of these two groups of hypertensive patients with "controlled" asleep SBP mean). According to this prospective evaluation, the asleep SBP mean, but not the daytime OBPM or the awake ambulatory BP mean, is the most significant and independent prognostic marker of CVD outcome.

On the basis of new evidence on the relationship between achieved OBPM and the risk of CVD morbidity and mortality documented in the SPRINT trial, the recent 2017 guidelines of the American College of Cardiology (ACC) and the American Heart Association (AHA) have established lower values of 130/80 mmHg for clinic SBP/DBP as new diagnostic thresholds for hypertension and therapeutic targets for treatment of all individuals aged ≥18 years regardless of age, sex, or concomitant complications including presence of diabetes, CKD, or history of past CVD event. According to these guidelines, the new proposed ABPM thresholds for diagnosis of hypertension in adults are 130/80 and 110/65 mmHg for the awake and asleep SBP/DBP means, respectively. However, the ACC/AHA guidelines do not provide any scientific evidence documenting neither the equivalence between these ABPM thresholds and the 130/80 mmHg cut-off values for OBPM nor the potential improved CVD event-free survival time of the proposed more intensive control of ambulatory BP.

All the results described above, including the main findings of the MAPEC and Hygia trials pertaining to the greater prognostic value of ABPM than OBPM, are derived from observational prospective studies consistently documenting that therapeutic BP targets in hypertensive individuals, i.e., persons at increased CVD risk, should be established in terms of proper control of asleep BP. To date, no prospective randomized study has ever before evaluated which should be the adequate therapeutic ABPM target for most effective reduction of CVD risk. Accordingly, the Tratamiento de Hipertensión Arterial Durante el Sueño study (THADEUS, i.e., Treatment of Hypertension During Sleep) has been designed to prospectively evaluate if the "intensive control" of asleep SBP mean proposed by the new ACC/AHA guidelines (<110 mmHg) in more effective than the so far "conventional control" (<120 mmHg) to reduce CVD morbidity and mortality in hypertensive individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 years.
2. All participants must: (i) have at randomization sleep-time hypertension according to the current ESH/ESC guidelines, i.e., asleep SBP mean ≥120 mmHg;1 (ii) adhere to a routine of daytime activity and nighttime sleep; and (iii) provide their written informed consent to participate into the study.

Exclusion Criteria:

1. Pregnancy.
2. History of drug/alcohol abuse within the last two years.
3. Night/shift-work employment.
4. Previous history of a systemic autoimmune disease or AIDS.
5. Evidence of a secondary form of hypertension, including coarctation of the aorta, hyperaldosteronism, renal artery stenosis, or pheochromocytoma
6. CVD disorders (unstable angina pectoris, heart failure, life-threatening arrhythmia, atrial fibrillation, kidney failure, and grade III-IV retinopathy). Previous CVD events will not be exclusionary if full physical and work activities are maintained.
7. Any surgical or medical condition which might alter the absorption, distribution, metabolism, or excretion of any drug, or, at the discretion of the investigator, might place the subject at higher risk from his/her participation in the study, or are likely to prevent the subject from complying with the requirements of the study or completing the trial period.
8. History of malignancy including leukemia and lymphoma (but not basal cell skin cancer), or any other severe, life-threatening disease within the past five years.
9. Inability to communicate and comply with all study requirements.
10. Intolerance to ABPM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5320 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular events | Median follow-up of 5 years
  Rate of cardiovascular events and stroke
New-onset type 2 diabetes | Median follow-up of 5 years
  Development of type 2 diabetes
New-onset CKD | Median follow-up of 5 years
  Development of chronic kidney disease

SECONDARY OUTCOMES:
Coronary events | Median follow-up of 5 years
  Rate of coronary events registered during follow-up
Cardiac events | Median follow-up of 5 years
  Rate of cardiac events registered during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, PhD, Principal Investigator — University of Vigo
Locations (9):
- Spain (9):
  - Complexo Hospitalario Universitario de Ourense, Ourense, Orense
  - CS A Estrada, A Estrada, Pontevedra
  - CS Panxón, Nigrán, Pontevedra
  - Centro de Salud de A Doblada, Vigo, Pontevedra
  - Centro de Salud de Bembrive, Vigo, Pontevedra
  - Centro de Salud de Sardoma, Vigo, Pontevedra
  - CS Teis, Vigo, Pontevedra
  - Bioengineering & Chronobilogy Labs., University of Vigo, Vigo, Pontevedra
  - CS San Roque, Vilagarcía de Arousa, Pontevedra

IPD SHARING:
Plan to Share IPD: Undecided